CLINICAL TRIAL: NCT01946178
Title: Clinical Study of a Focused Ultrasound Device for Treating Uterine Fibroids and Menorrhagia
Brief Title: Clinical Study of the Mirabilis High-Intensity Focused Ultrasound System for Non-Invasive Treatment of Uterine Fibroids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mirabilis Medica, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: No. 1006
Record Dates: First submitted 2013-09-16; First posted 2013-09-19 (Estimated); Results first posted 2016-03-25 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Uterine Fibroids (Leiomyomas)
Keywords: Uterine Fibroids; Leiomyomas; High-Intensity Focused Ultrasound Ablation; Ultrasonography
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Focused ultrasound treatment (Experimental): Patients in this arm will receive fibroid treatment using the Mirabilis High-Intensity Focused Ultrasound Treatment System.
  Interventions: Device: Mirabilis High-Intensity Focused Ultrasound Treatment System

INTERVENTIONS:
Device: Mirabilis High-Intensity Focused Ultrasound Treatment System — The intervention consists of a treatment session with the device, during which focused ultrasound energy is applied across the intact abdominal wall to ablate appropriately selected uterine fibroids under ultrasound imaging guidance.

SUMMARY:
The Mirabilis High-Intensity Focused Ultrasound (HIFU) Treatment System delivers therapeutic focused ultrasound energy to the uterus under integrated ultrasound imaging guidance to offer non-invasive treatment for uterine fibroids. The purpose of this clinical study is to assess the initial safety and performance of the Mirabilis HIFU Treatment System for transabdominal treatment of uterine fibroids in eligible women who are scheduled to undergo hysterectomy following treatment with the device or who are seeking relief from fibroid-related symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18-55 years
* Patients seeking relief from uterine fibroid related symptoms, including those scheduled to undergo abdominal hysterectomy due to benign pathology
* Patients able and willing to provide informed consent

Exclusion Criteria:

* Visible scar within the HIFU beam path that cannot be avoided
* Known or suspected abdominal adhesions between the anterior uterine serosa and the abdominal wall
* Currently pregnant or desire to become pregnant in the future
* Pelvic malignancy
* Pelvic congenital malformation
* Acute pelvic infection
* Otherwise determined by a physician to be inappropriate for the study

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2011-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lau, M.D., Study Director — Mirabilis Medica, Inc.
Locations (2):
- Mexico (2):
  - Hospital Torre Medica, Mexico City, Mexico City
  - Hospital Universitario, Universidad Autonoma de Nuevo Leon, Monterrey, Nuevo León

REFERENCES:
- [Result] Parsons JE, Lau MPH, Martin PJ, Islas Lagos JJ, Aguilar Aguirre JM, Garza Leal JG. Pilot Study of the Mirabilis System Prototype for Rapid Noninvasive Uterine Myoma Treatment Using an Ultrasound-Guided Volumetric Shell Ablation Technique. J Minim Invasive Gynecol. 2017 May-Jun;24(4):579-591. doi: 10.1016/j.jmig.2017.01.010. Epub 2017 Jan 18. PMID 28109895
- [Result] Garza Leal JG, Hernandez Leon I, Castillo Saenz L, Aguilar Aguirre JM, Islas Lagos JJ, Parsons JE, Darlington GP, and Lau MPH. In-Office Rapid Volumetric Ablation of Uterine Fibroids under Ultrasound Imaging Guidance: Preclinical and Early Clinical Experience with the Mirabilis Transabdominal HIFU Treatment System. Proceedings of the 14th International Symposium on Therapeutic Ultrasound. AIP Conference Proceedings 1821: 020001 (2017).
- [Result] Garza Leal JG, Hernandez Leon I, Castillo Saenz L, Aguilar Aguirre JM, Islas Lagos JJ, Parsons JE, Martin PM, and Lau MPH. Refinement of the Shell Ablation Technique for Rapid In-Office Treatment of Uterine Fibroids under Ultrasound Imaging Guidance using the Mirabilis Transabdominal HIFU System. 15th International Symposium on Therapeutic Ultrasound Program and Abstracts: 156 (2015).
- [Result] Lau M, Aguilar Aguirre JM, Islas Lagos JJ, and Garza Leal JG. Office Based High-Speed Ultrasound Image Guided HIFU (High Intensity Focused Ultrasound) Ablation of Uterine Fibroids. Gynecol. Surg. 11 (Suppl. 1): 149-150 (2014).
- [Result] Garza Leal JG, Hernandez Leon I, Castillo Saenz L, Aguilar Aguirre JM, Islas Lagos JJ, Parsons JE, Darlington GP, and Lau MPH. In-Office Rapid Volumetric Ablation of Uterine Fibroids under Ultrasound Imaging Guidance: Preclinical and Early Clinical Experience with the Mirabilis Transabdominal HIFU Treatment System. 14th International Symposium on Therapeutic Ultrasound Program and Abstracts: 43 (2014).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients underwent transabdominal uterine fibroid treatment with the Mirabilis High-Intensity Focused Ultrasound Treatment System between January 8, 2011 and November 21, 2014 at two clinical sites in Mexico. The study was completed on May 20, 2015.
Pre-assignment Details: Patients were screened prior to treatment for eligibility criteria including size, location, and tissue characteristics of their uterine fibroid(s). Those patients meeting the established eligibility criteria were then scheduled for treatment.
Groups:
- All Treated Patients: All patients who underwent treatment with the device
Period: Overall Study
Arm/Group | All Treated Patients
Started | 73
Completed | 71
Not Completed | 2
Not completed — Pregnancy | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported for the entire study population (all treated patients).
Arm/Group | All Treated Patients
Number analyzed (Participants) | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 73
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 42.8 [29 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73
  Male | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 73

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of All Adverse Events Encountered
Description: Safety of the treatment was determined by evaluating the incidence of Adverse Events and Adverse Device Effects. Adverse Device Effects are Adverse Events that are related to treatment with the device. Relatedness of an Adverse Event to the treatment was determined on a case-by-case basis by the investigator. The average number of Serious Adverse Device Effects per patient and the average number of Non-Serious Adverse Device Effects per patient are reported to provide numeric outcomes of this evaluation.
Time Frame: Adverse Events were monitored until the patient's exit from the study (up to 6 months post-treatment).
Population: All Adverse Device Effects are reported for the entire study population (all treated patients).
Measure: Mean (Full Range); unit: Adverse Device Effects / patient
Arm/Group | All Treated Patients
Number analyzed (Participants) | 73
Adverse Device Effects / patient
  Serious Adverse Device Effects Per Patient | 0 [0 to 0]
  Non-Serious Adverse Device Effects Per Patient | 0.95 [0 to 3]

2. Secondary Outcome: HIFU-related Non-Perfused Volume (NPV)
Description: Efficacy of the treatment was quantified by measuring the HIFU-related Non-Perfused Volume (NPV) of tissue in each patient using either post-treatment contrast-enhanced magnetic resonance imaging (MRI) or pathology assessment following hysterectomy. The NPV is used to measure the amount of tissue that was treated during the procedure.
Time Frame: The NPV was measured between 0 and 7 days post-treatment.
Population: HIFU-related Non-Perfused Volumes (NPVs) are reported for all treated patients in whom they were observed following treatment. NPV outcomes are stratified between two cohorts: an early Development Cohort and a final Validation Cohort.
Measure: Mean (Full Range); unit: cubic centimeters (cc)
Groups:
- Development Cohort With NPVs Observed: The Development Cohort includes the first 37 patients treated in the study sequence. Treatments in the Development Cohort were used for dose-ranging purposes to develop the most appropriate HIFU parameters for uterine fibroid treatment with the device. Outcomes are reported for the 33 out of 37 patients (89.2%) in the Development Cohort with NPVs observed following treatment.
  Overall, 68 out of 73 patients (93.2%) in the entire study had NPVs observed following treatment.
- Validation Cohort With NPVs Observed: The Validation Cohort includes the last 36 patients treated in the study sequence. Treatments in the Validation Cohort were used to refine and validate the final HIFU parameters for uterine fibroid treatment with the device. Outcomes are reported for the 35 out of 36 patients (97.2%) in the Validation Cohort with NPVs observed following treatment.
  Overall, 68 out of 73 patients (93.2%) in the entire study had NPVs observed following treatment.
Arm/Group | Development Cohort With NPVs Observed | Validation Cohort With NPVs Observed
Number analyzed (Participants) | 33 | 35
cubic centimeters (cc) | 20.1 [0.6 to 123.0] | 46.1 [1.1 to 284.7]

3. Post Hoc Outcome: Total Time Required to Deliver Treatment
Description: The total treatment time was measured for each patient from the beginning of HIFU energy emission until HIFU energy emission stopped.
Time Frame: The total treatment time was measured on the day of treatment.
Population: Total treatment times are reported for all treated patients. Total treatment times are stratified between two cohorts: an early Development Cohort and a final Validation Cohort.
Measure: Mean (Full Range); unit: minutes
Groups:
- Entire Development Cohort: The Development Cohort includes the first 37 patients treated in the study sequence. Treatments in the Development Cohort were used for dose-ranging purposes to develop the most appropriate HIFU parameters for uterine fibroid treatment with the device. Outcomes are reported for all 37 patients in the Development Cohort.
- Entire Validation Cohort: The Validation Cohort includes the last 36 patients treated in the study sequence. Treatments in the Validation Cohort were used to refine and validate the final HIFU parameters for uterine fibroid treatment with the device. Outcomes are reported for all 36 patients in the Validation Cohort.
Arm/Group | Entire Development Cohort | Entire Validation Cohort
Number analyzed (Participants) | 37 | 36
minutes | 4.9 [1.1 to 11.3] | 3.6 [1.5 to 9.5]

ADVERSE EVENTS:
Time Frame: Monitoring for Adverse Events occurred from January 8, 2011 until May 20, 2015. Adverse Events were monitored until each patient's exit from the study, which was up to 6 months following treatment.
Description: All Adverse Events are reported for all patients receiving treatment, including those events not related to treatment. Adverse Events were reported spontaneously by patients, observed by the investigator or other personnel, and/or elicited during patient queries at regular follow-up intervals. Descriptions were mapped to standardized terms.
Arm/Group | All Treated Patients
Serious Adverse Events (participants affected / at risk) | 2/73
Other Adverse Events (participants affected / at risk) | 53/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Treated Patients (N=73)
Diarrhea unrelated to treatment (General disorders) | 1 (1) — related to concurrent E. coli infection
Depressed respiration with apnea unrelated to treatment (General disorders) | 1 (1) — related to analgesic administration
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Treated Patients (N=73)
Abdominal cramping pain during HIFU (General disorders) | 42 (46)
Abdominal cramping pain post HIFU (General disorders) | 14 (16)
Vaginal bleeding (General disorders) | 7 (7)
Nausea with vomiting unrelated to treatment (General disorders) | 4 (4)
Headache unrelated to treatment (General disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days